CLINICAL TRIAL: NCT05841121
Title: Antenatal Dexamethasone for Late Preterm Deliveries: a Randomized Controlled Trial
Brief Title: Antenatal Dexamethasone for Late Preterm Deliveries
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Chau Hoang Minh Le, Principal Investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 49/2566
Record Dates: First submitted 2023-04-03; First posted 2023-05-03 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Distress of Newborn; Preterm Birth
Keywords: Late preterm infants; Respiratory distress
MeSH Terms: conditions — Pulmonary Atelectasis; Premature Birth; Dyspnea | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Participants are women with singleton pregnancy, from 18 to 45 years old, at 34+0/7 to 36+6/7 weeks of gestation and at high risk for delivery during the late preterm period in the next 7 days.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone group (Experimental): The intervention is antenatal dexamethasone. Participants in the intervention group will be given a course of four intramuscular injections of dexamethasone 6 mg (1.2 milliliter), 12 hours apart.
  Interventions: Drug: Dexamethasone
- Control group (No Intervention): Participants in the control group will be received standard care.

INTERVENTIONS:
Drug: Dexamethasone — Antenatal dexamethasone will be given a course of four intramuscular injections of dexamethasone 6 mg (1.2 milliliter), 12 hours apart.
  Arms: Dexamethasone group

SUMMARY:
The goal of this clinical trial is to compare dexamethasone in late preterm deliveries. The main questions it aims to answer are: Does antenatal dexamethasone reduce the need for respiratory support in late preterm infants? Does antenatal dexamethasone reduce neonatal morbidities and mortality? Does antenatal dexamethasone reduce admission to Neonatal Intensive Care Unit and length of hospital stay? Participants will be allocated into 2 groups: intervention with dexamethasone IM and control (standard care). Investigators will compare these two groups to see if antenatal dexamethasone reduces the need for respiratory support in late preterm infants, neonatal morbidities and mortality, admission to NICU and length of hospital stay.

DETAILED DESCRIPTION:
Study design: The study is a double-blinded randomized controlled trial, parallel group. The sequence of randomization will be generated by using an online tool (https://www.sealedenvelope.com/simple-randomiser/v1/lists) with 2 groups of treatments with ratio 1:1, block of variable size (2,4,6), list length 302, no stratification. After having a randomization sequence, the symbol of group (control or intervention) will be kept in a sealed envelope. These envelops will be also put in the order as the allocation sequence. Assessors and investigators will be blinded to the group allocation.

Participants: Participants are women with singleton pregnancy, from 18 to 45 years old, at 34+0/7 to 36+6/7 weeks of gestation and at high risk for delivery during the late preterm period in the next 7 days.

Intervention: Antenatal dexamethasone. Participants in the intervention group will be given a course of four intramuscular injections of dexamethasone 6 mg (1.2 milliliter), 12 hours apart.

Comparison: Standard care. Outcomes: Primary outcome: Need for any respiratory support in first 72 hours, which is determined when babies need to be supported with continuous positive airway pressure (CPAP), high-flow nasal cannula (HFNC), supplemental oxygen, or mechanical ventilation in first 72 hours to keep the saturation in a proper range (90-95%).

Sample size is 300 participants in 2 groups: intervention group and control group.

Place: The study will be conducted at Danang Hospital for Women and Children, Danang, Vietnam.

Eligibility of participants will be assessed at admission area of delivery department. One senior obstetrician will introduce the study to the patient by using the study information sheet. If the pregnant woman agrees to join in the research, the writen consent will be delivered to her and she will sign on it. When participants agrees, one sealed envelope with a number inside will be opened to allocate which group she involves. At that time, Eligibility criteria and Part 1 of the CRF will also be filled.

After randomization, pregnant women will be monitored at delivery rooms until delivery or c-section. After birth, both mother and baby will be closed monitored and assessed until transferred to post-natal wards or neonatal unit. Part 2. Labour and at birth Part 3. Newborn outcomes Part 4: Maternal outcomes will be collected.

If infants discharge before 28 days old, the follow-up section will be done at follow-up clinic of neonatal unit. Information about outcome (alive or death), any re-admission to hospital (number of time and reasons), and nutrition (types of milk (breast milk, formula milk or mix), feeding methods (breast feeding, bottle, tube/cup/spoon) will be collected for Part 5 of CRF.

ELIGIBILITY:
Inclusion Criteria:

* 34+0/7 to 36+6/7 weeks
* Expected preterm delivery for any indications in the next 7 days.

Exclusion Criteria:

* Fetal death
* Severe fetal malformation
* Twin or multiple pregnancy
* Maternal contraindication to dexamethasone: hypersensitive with steroids, any infection
* Severe maternal conditions such as eclampsia, cardiac arrest, antepartum hemorrhage due to placenta previa or abruption
* Delivery estimated within 2 hours: total cervical dilation
* Received steroids within 1 week

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 294 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of respiratory support | First 72 hours of life
  Rate of babies requiring any respiratory support such as continuous positive airway pressure (CPAP), high-flow nasal cannula (HFNC), supplemental oxygen, or mechanical ventilation in first 72 hours to keep the saturation in a proper range (90-95%).

SECONDARY OUTCOMES:
Neonatal respiratory morbidities | From birth to 28 days of life or death
  Rate of respiratory morbidities: RDS, TTN, Surfactant administration, Need for mechanical ventilation, Apnea, BPD
Neonatal co-morbidities | From birth to 28 days of life or death
  Rate of co-morbidities: resuscitation after birth, other morbidities: Hypoglycemia, Hypothermia, Early onset infection, Late onset infection, Jaundice need phototherapy, IVH, NEC, Admission to NICU, Neonatal mortality; average hospital days
Neonatal treatment outcomes | From birth to 28 days of life or death
  Rate of admission to NICU, Neonatal mortality rate, average hospital days
Maternal secondary outcomes | First week after delievery
  Rate of maternal post-partum infection, rate of c-section
Maternal outcomes | First week after delievery
  Average hospital days

CONTACTS AND LOCATIONS:
Locations (1):
- Danang HOspital for Women and Children, Da Nang, Vietnam

REFERENCES:
- [Derived] Le CHM, Tran HT, Huynh QK, Chaithongwongwatthana S. Impact of Antenatal Dexamethasone on Respiratory Outcomes in Late Preterm Infants in a Vietnamese Tertiary Hospital: A Randomised Controlled Trial. Acta Paediatr. 2025 Dec 26. doi: 10.1111/apa.70417. Online ahead of print. PMID 41452963